CLINICAL TRIAL: NCT01156441
Title: Medical Versus Surgical Management of Patients With Moderate Mitral Regurgitation Following Percutaneous Coronary Intervention for Myocardial Infarction: A Pilot Prospective Randomized Trial
Brief Title: Medical Versus Surgical Management of Moderate Mitral Regurgitation Following Percutaneous Coronary Intervention
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAS-SIU-10-003-1
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Myocardial Infarction; Mitral Regurgitation
Keywords: Myocardial Infarction; Mitral Regurgitation; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction; Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgical mitral valve repair (Experimental): Non-invasive transesophageal echocardiography will be performed on all study volunteers to determine if the individual has mitral regurgitation and, if so, to what degree. Mitral valve repair will be performed with mitral valve annuloplasty via median sternotomy, utilizing cardiopulmonary bypass and moderate hypothermia.
  Interventions: Procedure: surgical mitral valve repair w/ mitral valve annuloplasty
- control: medical management (No Intervention): Clinical observation will be continued without surgery. Non-invasive transesophageal echocardiography will be performed on all study volunteers to determine if the individual has mitral regurgitation and, if so, to what degree.

INTERVENTIONS:
Procedure: surgical mitral valve repair w/ mitral valve annuloplasty — Mitral valve repair will be performed via median sternotomy, utilizing cardiopulmonary bypass and moderate hypothermia. The mitral valve will be approached through a left atrial incision. Following inspection of the valve, mitral valve annuloplasty will be accomplished with a complete semi-rigid annuloplasty ring. Additional techniques to address residual regurgitation will be at the discretion of the surgeon. The left atriotomy will then be closed and the patient weaned off and separated from the cardiopulmonary bypass.
  Intraoperative transesophageal echocardiography will be performed on all study volunteers.
  Other Names: mitral valve annuloplasty
  Arms: surgical mitral valve repair

SUMMARY:
The pilot prospective randomized trial is designed to determine the safety and feasibility of enrolling patients to surgically correct residual Mitral Regurgitation (MR) following Percutaneous Coronary Intervention (PCI) for Myocardial Infarction (MI) verses ongoing medical management of MR. The investigators hypothesize that if moderate MR is corrected in this patient subset, the patients will have improved outcomes as measured by decreased number of major adverse cardiac events, including death, congestive heart failure requiring hospitalization, atrial fibrillation, deterioration of New York Heart Association (NYHA) functional status and improved quality of life.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) is a frequent complication of myocardial infarction. Ischemic MR portends a poor prognosis on long term follow up. This pilot prospective randomized trial is a safety and feasibility trial to evaluate mitral valve repair versus surgical management in patients with residual MR after primary percutaneous coronary intervention (PCI). Patients will be screened for possible inclusion to identify those that have first MI treated with primary PCI. Patients with moderate MR at 6 or more weeks following first primary PCI will be randomized to continued medical management versus surgical mitral valve repair. Patients with previous or subsequent coronary artery bypass surgery and patients with severe ventricular dysfunction will be excluded. Patients will be followed for one year from the time of randomization. The safety and feasibility data will be used to design a large trial powered to detect a difference in mortality between treatment arms.

Results of this study could lead to a radical change in the treatment paradigm for patients with ischemic MR following PCI for acute MI. In addition, insight gained from this study could advance our understanding of the interrelationship between LV remodeling and MR and shed some light into the mechanism of ventricular function deterioration following MI. Moreover, it may provide a framework for the development of further recommendations with respect to the indications for surgical intervention in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone PCI for first acute MI (index MI) since 7/1/09 at MMC and STJ
* documented moderate mitral regurgitation on follow up echocardiography six or more weeks after PCI procedure
* English speaking

Exclusion Criteria:

* CABG after PCI for acute MI
* History of previous MI prior to index MI
* History of previous PCI or CABG prior to index PCI
* EF <30 % on the echocardiogram at 6 weeks after PCI for MI

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
patient survival | baseline to 1 year
  Patient survival will be prospectively documented for all study subjects from recruitment through one year. A stopping rule for the surgical arm is a pre-specified cut-off of 5% based on the method proposed by Kramar and Bascoul-Mollevi in "Early Stopping Rules in Clinical Trials Based on Sequential Monitoring of Serious Adverse Events" [39]. A data and safety monitoring board (DSMB) that includes five independent investigators and a statistician has been established to conduct ongoing study review to maintain safety of all participants.

SECONDARY OUTCOMES:
congestive heart failure requiring hospitalization | baseline and 1 year
  Hospitalization for congestive heart failure will be prospectively documented for all study subjects from recruitment through one year.
mitral regurgitation grade | baseline and 1 year
  Transthoracic echocardiogram will be obtained to assess the presence and or severity of mitral regurgiation.
new atrial fibrillation | baseline, 3 months, 6 months and 1 year
  EKG will be obtained during routine clinical follow up visits and at one year.
NYHA functional class | baseline, 3 months, 6 months and 1 year
  This will be assessed via patient questionnaire using the standard NYHA classification.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Vassileva, M.D., Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Vassileva CM, Boley T, Markwell S, Hazelrigg S. Meta-analysis of short-term and long-term survival following repair versus replacement for ischemic mitral regurgitation. Eur J Cardiothorac Surg. 2011 Mar;39(3):295-303. doi: 10.1016/j.ejcts.2010.06.034. Epub 2010 Aug 19. PMID 20727782
- See also: Southern Illinois University School of Medicine website — http://www.siumed.edu